CLINICAL TRIAL: NCT04771819
Title: Safety and Performance of SoftOx Wound Irrigation Solution (SWIS) Compared to Normal Saline (NS) in Human Experimental Suction Blister Wounds
Brief Title: Safety and Performance of SWIS in Superficial Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SoftOx Solutions AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SWIS-02
Record Dates: First submitted 2020-11-23; First posted 2021-02-25 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Wound of Skin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SoftOx Wound Irrigation Solution (SWIS) (Experimental): Blister wounds will be irrigated and soaked for 15 minutes.
  Interventions: Device: SWIS
- Normal Saline (Active Comparator): Blister wounds will be irrigated and soaked for 15 minutes.
  Interventions: Device: SWIS

INTERVENTIONS:
Device: SWIS — Bilateral experimental blister wounds on each forearm. The wound on one arm is rinsed with experimental solution (SWIS) and the contralateral wound on the other arm is rinsed With Saline as a comparator.

SUMMARY:
This is an open, evaluator blinded, intra-comparative, randomized, non-inferiority investigation prior to CE mark to confirm safety and performance of the SWIS device when used as intended, i.e. as an irrigation solution for mechanical rinsing of breached or compromised skin as a result from acute wounds.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and intact skin where the blister suction wounds will be induced
* Been informed of the nature, the scope and the relevance of the clinical investigation
* Voluntarily agreed to participation and has duly signed the Information Consent Form

Exclusion Criteria:

1. Participating in any other clinical investigation
2. Disease that may interfere with the wound healing, e.g. diabetes, arterial-, renal-, liver, or cardiac insufficiency, chronic obstructive lung disease, cancer, autoimmune disease, edema of the arm, severe obesity, severe psychiatric disease, dementia or previous known wound healing problems, as judged by the investigator
3. Active skin disease, e.g. dermatitis, psoriasis and wounds, and/or tattoos in the areas where suction blister wounds will be induced, as judged by the investigator
4. Daily smoker
5. Pregnancy
6. Systemic immunosuppressive treatment
7. Uncontrolled pain that may interfere with the investigation outcome, as judged by the investigator
8. Allergy to hypochlorous acid, acetic acid or any other remedies/material used in the clinical investigation
9. Not able to read or understand Danish
10. Any other conditions that as judged by the investigator may make follow-up or investigation inappropriate
11. That according to the Declaration of Helsinki is deemed unsuitable for study enrolment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Degree (percentage) re-epithelialization in the suction blister wound on day 10 in the SWIS treated wound versus NS treated wound | From baseline to day 10
  Measure the degree of re-epithelialization to evaluate any differences between the treatments.

SECONDARY OUTCOMES:
Degree (percentage) re-epithelialization in the suction blister wound on day 4 in the SWIS treated wound versus NS treated wound. | From baseline to day 4
  Evaluate any differences between the two treatments on early epithelialization.
Percentage of suction blister wounds healed on day 10 in the SWIS treated wound versus NS treated wound | Day 10
  Evaluate any differences between the two treatments on day 10
Percentage of suction blister wounds healed on day 17 (+/- 1 day) in the SWIS treated wound versus NS treated wound | Day 17
  Evaluate any differences between the two treatments on day 17
Percentage of suction blister wounds with >30% CFU reduction in the SWIS treated wound and NS treated wound respectively if positive CFU level prior irrigation | Day 4
  Evaluate any differences between the two treatments on reducing bacterial load in wounds
Subject evaluation of pain during each irrigation procedure on days 0, 2 and 4 in the SWIS treated wound versus NS treated wound | Baseline (day 0), day 2 and day 4
  Evaluate any differences on pain using VAS scale between the SWIS and Normal Saline during irrigation and moistening on day 0,2 and 4.
The incidence and severity of adverse events | Baseline to day 17
  Evaluate any differences between the two treatments regarding side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No